CLINICAL TRIAL: NCT01424839
Title: SIOP CNS GCT II: Prospective Trial for the Diagnosis and Treatment of Children, Adolescents and Young Adults With Intracranial Germ Cell Tumors
Brief Title: Prospective Trial for the Diagnosis and Treatment of Intracranial Germ Cell Tumors
Acronym: SIOPCNSGCTII
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Muenster (Other)
Collaborators: Deutsche Kinderkrebsstiftung (Other); Hannover Medical School (Other); German Society for Pediatric Oncology and Hematology GPOH gGmbH (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UKM08_0057; 2009-018072-33 (EudraCT Number)
Record Dates: First submitted 2011-08-11; First posted 2011-08-29 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Intracranial Germ Cell Tumors
Keywords: SIOP CNS GCT II; Patients with the primary disease of an Intracranial Germ Cell Tumors
MeSH Terms: interventions — Craniospinal Irradiation; Ice; Cisplatin; Etoposide; Ifosfamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Germinoma metastatic (Other): • Metastatic or incompletely staged germinomas (± teratoma) Do not receive chemotherapy in this protocol
  Radiotherapy
  * Metastatic or incompletely staged pure germinoma 24 Gy (15 fractions) to craniospinal axis with a 16 Gy (10 fraction) boost to tumour bed and any intracranial metastases and spinal deposits (total tumour dose 40 Gy)
  * Metastatic germinoma plus teratoma (incompletely resected) 24 Gy (15 fractions) to craniospinal axis ; 30.4 Gy (19 fraction) boost to tumour bed and 16 Gy (10 frac-tion) boost to metastases (total tumour dose 54.4 Gy)
  Interventions: Radiation: craniospinal irradiation
- germinoma non-metastatic (Other): Chemotherapy:
  • Non-metastatic fully staged germinoma (± teratoma) Two courses (1 and 3) of Etoposide and Carboplatin, alternating with two courses (2 and 4) of Etoposide and Ifosfamide Note: Bifocal germinoma (pineal+suprasellar) are treated as non-metastatic germinoma, if staging shows no additional dissemination
  Radiotherapy
  * Non-metastatic pure germinoma in PR/SD After Chemotherapy: 24 Gy (15 fractions) to whole ventricles with a 16 Gy (10 fraction) boost to tumour bed (total tumour dose 40 Gy)
  * Non-metastatic germinoma in CR After Chemotherapy: 24 Gy (15 fractions) to whole ventricles
  * Non-metastatic germinoma plus teratoma (incompletely resected) After Chemotherapy: 24 Gy (15 fractions) to whole ventricles; 30.4 Gy (19 fraction) boost to tumour bed (total tumour dose 54.4 Gy)
  Interventions: Drug: Carboplatin, Etoposide, Ifosfamide; Radiation: ventricular irradiation
- Non-germinoma non-metastatic standard risk (Other): Chemotherapy:
  • Standard risk non-germinomatous malignant GCT Four courses of Etoposide, Cisplatin and Ifosfamide (standard treatment ) After Chemotherapy: 54 Gy focal radiotherapy in 30 fractions
  Interventions: Drug: Cisplatin, etoposide, Ifosfamide (standard); Radiation: focal irradiation
- Non-Germinoma metastatic standard risk (Other): Chemotherapy Four courses of Etoposide, Cisplatin and Ifosfamide (standard treatment ) Radiotherapy After Chemotherapy: 30 Gy (20 fractions) to craniospinal axis with 24 Gy (15 fraction) boosts to tumour site and any intracranial metastases (total tumour dose 54 Gy) and 20.8 Gy (13 fraction) boosts to spinal deposits (total dose 50.8 Gy)
  Interventions: Radiation: craniospinal irradiation; Drug: Cisplatin, etoposide, Ifosfamide (standard)
- Non-germinoma non-metastatic high risk (Other): Chemotherapy Two courses of standard Etoposide, Cisplatin and Ifosfamide, followed by two dose intensified courses of Etoposide, Cisplatin and Ifosfamide with stem cell support Radiotherapy After Chemotherapy: 54 Gy focal radiotherapy in 30 fractions
  Interventions: Drug: Cisplatin, Etoposide, Ifosfamide (high dose); Radiation: focal irradiation
- Non-Germinoma metastatic high risk (Other): Chemotherapy Two courses of standard Etoposide, Cisplatin and Ifosfamide, followed by two dose intensified courses of Etoposide, Cisplatin and Ifosfamide with stem cell support Radiotherapy After Chemotherapy: 30 Gy (20 fractions) to craniospinal axis with 24 Gy (15 fraction) boosts to tumour site and any intracranial metastases (total tumour dose 54 Gy) and 20.8 Gy (13 fraction) boosts to spinal deposits (total dose 50.8 Gy)
  Interventions: Radiation: craniospinal irradiation; Drug: Cisplatin, Etoposide, Ifosfamide (high dose)
- Teratoma (No Intervention): collection of information on surgery, applied treatment and outcome

INTERVENTIONS:
Radiation: craniospinal irradiation — * Metastatic or incompletely staged pure germinoma 24 Gy (15 fractions) to craniospinal axis with a 16 Gy (10 fraction) boost to tumour bed and any intracra-nial metastases and spinal deposits (total tumour dose 40 Gy)
  * Metastatic germinoma plus teratoma (incompletely resected) 24 Gy (15 fractions) to craniospinal axis ; 30.4 Gy (19 fraction) boost to tumour bed and 16 Gy (10 frac-tion) boost to metastases (total tumour dose 54.4 Gy)
  * Patients with metastastic non-germinomatous disease at diagnosis After Chemotherapy: 30 Gy (20 fractions) to cranio-spinal axis with 24 Gy (15 fraction) boosts to tumour site and any intracranial metastases (total tumour dose 54 Gy) and 20.8 Gy (13 fraction) boosts to spinal deposits (total dose 50.8 Gy)
  Arms: Germinoma metastatic; Non-Germinoma metastatic high risk; Non-Germinoma metastatic standard risk
Drug: Carboplatin, Etoposide, Ifosfamide — • Non-metastatic fully staged germinoma (± teratoma) Two courses (1 and 3) of Etoposide and Carboplatin, alternating with two courses (2 and 4) of Etoposide and Ifosfamide
  Arms: germinoma non-metastatic
Radiation: ventricular irradiation — * Non-metastatic pure germinoma in PR/SD After Chemotherapy: 24 Gy (15 fractions) to whole ventricles with a 16 Gy (10 fraction) boost to tumour bed (total tumour dose 40 Gy)
  * Non-metastatic germinoma in CR After Chemotherapy: 24 Gy (15 fractions) to whole ventricles
  * Non-metastatic germinoma plus teratoma (incompletely resected) After Chemotherapy: 24 Gy (15 fractions) to whole ventricles; 30.4 Gy (19 fraction) boost to tumour bed (total tumour dose 54.4 Gy)
  Arms: germinoma non-metastatic
Drug: Cisplatin, etoposide, Ifosfamide (standard) — Four courses of Etoposide, Cisplatin and Ifosfamide (standard treatment )
  Arms: Non-Germinoma metastatic standard risk; Non-germinoma non-metastatic standard risk
Drug: Cisplatin, Etoposide, Ifosfamide (high dose) — Two courses of standard Etoposide, Cisplatin and Ifosfamide, followed by two dose intensified courses of Etoposide, Cisplatin and Ifosfamide with stem cell support
  Arms: Non-Germinoma metastatic high risk; Non-germinoma non-metastatic high risk
Radiation: focal irradiation — • Patients with localised non-germinomatous disease at diagnosis After Chemotherapy: 54 Gy focal radiotherapy in 30 fractions
  Arms: Non-germinoma non-metastatic high risk; Non-germinoma non-metastatic standard risk

SUMMARY:
STUDY DESIGN:

Prospective, non-randomised multicentre study with patients stratified according to risk groups INVESTIGATIONAL MEDICINAL PRODUCTS The IMPs on this trial are Carboplatin, Cisplatin, Ifosfamide and Etoposide (as approved by German competent authority).

PRIMARY OBJECTIVES:

Germinoma

* To maintain current high event-free survival (EFS) rates using a risk adapted approach
* In localised germinoma: to omit whole brain and spinal irradiation by using combined treatment with standard chemotherapy and ventricular irradiation (+/- boosts)
* In bifocal tumours (pineal + suprasellar): to treat as non-metastatic disease and to omit whole brain and spinal irradiation by using combined treatment with standard chemotherapy and ventricular irradiation (+/- boosts)
* In metastatic disease: to maintain current excellent EFS in metastatic germinoma with craniospinal irradiation Malignant non-germinoma

To improve EFS:

* by dose escalation of chemotherapy in patients identified as high risk at diagnosis ( age < 6 years and/or AFP serum / CSF > 1000 ng/ml)
* by standardising the surgical approach for residual disease after treatment Teratoma
* To register patients and collect data regarding diagnostics, treatment and outcome in order to develop future treatment strategies

SECONDARY OBJECTIVES:

Germinoma

* To minimise long term effects of irradiation by sparing spinal and whole brain radiotherapy in non-metastatic disease Malignant non-germinoma
* In standard risk to maintain EFS with chemotherapy and local irradiation Teratoma
* To evaluate the influence of surgery and treatment on outcome to assist in the development of a fu-ture treatment strategy For all histological subtypes
* To improve accuracy of diagnosis and staging in all registered patients
* To standardise neurosurgical intervention
* For all patients requiring biopsy or resection according to protocol guidelines, to collect and to store tumour material, and CSF where possible, for use in future biological studies.

ENDPOINTS / Criteria for evaluation:

Main end point

Event-free survival, defined as minimum time from the date of diagnosis to:

* Death from any cause
* Relapse
* Progressive disease on therapy
* Or second malignancy

Secondary end points

* Overall survival, defined as time to death from any cause, measured from the date of diagnosis
* Short and long term toxicity.

DETAILED DESCRIPTION:
PATIENT POPULATION Age of patients: no lower or upper age limit; Estimated number: 400 malignant germ cell tumours

Diagnosis and main criteria for inclusion/exclusion:

Intracranial Germ Cell tumours of any histology and intracranial site and dissemination

Inclusion criteria

* Main residence in one of the participating countries
* Primary diagnosis of an intracranial germ cell tumour
* Written consent for trial participation, treatment according to the protocol and consent for data trans-fer

Exclusion criteria:

* Tumour entity other than primary intracranial germ cell tumour or CNS GCT as second malignancy
* Primary diagnosis pre-dating the opening of SIOP CNS GCT II in the participating country of registration
* Medical, psychiatric or social conditions incompatible with trial treatment or treatment according to protocol is not intended
* Participation within a different trial for treatment of germ cell tumours and/or concurrent treatment within any other clinical trial. The only exceptions to this are trials with different endpoints, involving aspects of supportive treatment which can run parallel to SIOP CNS GCT II without influencing the outcome of this trial e.g. trials on antiemetics, antimycotics, antibiotics, strategies for psychosocial support etc.
* Pregnancy and lactation
* Any treatment not given according to protocol prior to registration

TREATMENT:

GERMINOMA

Chemotherapy:

* Non-metastatic fully staged germinoma (± teratoma) Two courses (1 and 3) of Etoposide and Carboplatin, alternating with two courses (2 and 4) of Etoposide and Ifosfamide Note: Bifocal germinoma (pineal+suprasellar) are treated as non-metastatic germinoma, if stag-ing shows no additional dissemination
* Metastatic or incompletely staged germinomas (± teratoma) Do not receive chemotherapy in this protocol

Radiotherapy:

* Non-metastatic pure germinoma in PR/SD After Chemotherapy: 24 Gy (15 fractions) to whole ventricles with a 16 Gy (10 fraction) boost to tumour bed (total tumour dose 40 Gy)
* Non-metastatic germinoma in CR After Chemotherapy: 24 Gy (15 fractions) to whole ventricles
* Metastatic or incompletely staged pure germinoma 24 Gy (15 fractions) to craniospinal axis with a 16 Gy (10 fraction) boost to tumour bed and any intracranial metastases and spinal deposits (total tumour dose 40 Gy)
* Non-metastatic germinoma plus teratoma (incompletely resected) After Chemotherapy: 24 Gy (15 fractions) to whole ventricles; 30.4 Gy (19 fraction) boost to tumour bed (total tumour dose 54.4 Gy)
* Metastatic germinoma plus teratoma (incompletely resected) 24 Gy (15 fractions) to craniospinal axis ; 30.4 Gy (19 fraction) boost to tumour bed and 16 Gy (10 frac-tion) boost to metastases (total tumour dose 54.4 Gy)

NON-GERMINOMA (± TERATOMA)

Chemotherapy:

* Standard risk non-germinomatous malignant GCT Four courses of Etoposide, Cisplatin and Ifosfamide (standard treatment )
* High risk non-germinomatous malignant GCT Two courses of standard Etoposide, Cisplatin and Ifosfamide, followed by two dose intensified courses of Etoposide, Cisplatin and Ifosfamide with stem cell support

Resection of residual tumour after 3 courses chemotherapy (if indicated), followed by: 4th course. If vi-able cells are found in the resected tumour specimen patient is transferred to the high risk arm

Radiotherapy for standard and high risk non-germinomatous malignant GCT:

* Patients with localised disease at diagnosis After Chemotherapy: 54 Gy focal radiotherapy in 30 fractions
* Patients with metastatic disease at diagnosis After Chemotherapy: 30 Gy (20 fractions) to craniospinal axis with 24 Gy (15 fraction) boosts to tumour site and any intracranial metastases (total tumour dose 54 Gy) and 20.8 Gy (13 fraction) boosts to spinal deposits (total dose 50.8 Gy)

SPECIAL ASPECTS:

Central response evaluation on a national basis:

Germinoma: In all patients with localised germinoma a central national radiological review is mandatory for response evaluation to chemotherapy and decision if only ventricular irradiation or an additional tu-mour boost has to be performed.

Non-Germinoma: After three courses of chemotherapy to evaluate response to treatment and to deter-mine necessity of surgery in case of residual before radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Main residence in one of the participating countries
* Primary diagnosis of an intracranial germ cell tumour
* Written consent for trial participation, treatment according to the protocol and consent for data transfer

Exclusion Criteria:

* Tumour entity other than primary intracranial germ cell tumour or CNS GCT as second malignancy
* Primary diagnosis pre-dating the opening of SIOP CNS GCT II in the participating country of registration
* Medical, psychiatric or social conditions incompatible with trial treatment or treatment according to protocol is not intended
* Participation within a different trial for treatment of germ cell tumours and/or concurrent treatment within any other clinical trial. The only exceptions to this are trials with different endpoints, involving aspects of supportive treatment which can run parallel to SIOP CNS GCT II without influencing the outcome of this trial e.g. trials on antiemetics, antimycotics, antibiotics, strategies for psychosocial support etc.
* Pregnancy and lactation
* Any treatment not given according to protocol prior to registration

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2011-10; Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
survival | 5 years event free survival
  Survival rates in respect to applied treatment , according to Kaplan-Meier estimation , 5 years event free survival

SECONDARY OUTCOMES:
short and long term toxicity | until 7 years after start of trial
  toxicity of treatment will be assessed with CTC criteria, severe toxicity will be analysed by safety desk
overall survival | 7 years after start of trial
  Overall survival will be measured by Kaplan -Meier Estimation , 5 years overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Calaminus, MD, Principal Investigator — University Hospital Muenster
Locations (1):
- University Hospital Muenster, Münster, Germany

REFERENCES:
- [Derived] Rajagopal R, Leong SH, Jawin V, Foo JC, Ahmad Bahuri NF, Mun KS, Azman RR, Loh J, Yap TY, Ariffin H, Moreira DC, Gottardo NG, Bouffet E, Ganesan D. Challenges in the Management of Childhood Intracranial Germ Cell Tumors in Middle-Income Countries: A 20-Year Retrospective Review From a Single Tertiary Center in Malaysia. J Pediatr Hematol Oncol. 2021 Oct 1;43(7):e913-e923. doi: 10.1097/MPH.0000000000002116. PMID 33633029